CLINICAL TRIAL: NCT01745406
Title: Benefits of the Involvement of Nurses in Meetings Between Physicians and the Families of Patients in the ICU.
Acronym: NEWS
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Fondation de France (Other); French Society for Intensive Care (Other)
Responsible Party: Sponsor
Other Study IDs: CPP/107-11
Record Dates: First submitted 2012-09-28; First posted 2012-12-10 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2013-04

CONDITIONS: Family Satisfaction; Healthcaregiver Satisfaction; Family PTSD; Family HADS; Family Traumatic Dissociation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Doctor and nurse
- Doctor without nurse

SUMMARY:
When a patient is admitted to the ICU this often happens so suddenly that this can create a significant amount of stress and anxiety for family members for several reasons. Firstly, the family does not have a pre existing relationship with the ICU team. Secondly, the urgency of the situation and the technic it requires is often such that minimal information can be given to family members. And finally, as a result of the unpredictability of each patient's condition, it can be difficult to predict outcome for family members. Together, these factors compound the stress and anxiety of family members. This anxiety is natural and it is important for health caregivers to be able to offer the best support possible. A high quality communication provided by structured information given by physicians and nurses as well could improve support to the families and lead to greater satisfaction.

Giving information to families during meetings is crucial at 3 moments: at the first day when the patient is admitted, at day 3, weekly and each time important news is given (surgery, deterioration in condition, end-of-life).

The purpose of this project is to evaluate if the involvement of nurses during those meetings could improve quality in communication which is assessed by mixed methods. Families and healthcare workers satisfaction will be assessed by qualitative methodology. Family peritraumatic stress, symptoms of anxiety and depression and PTSD will be assessed using validated scales.

Training of healthcare workers will be done by role play. Information to the families is delivered using a framework for physicians and nurses. All the meetings of the study will be audited by a psychologist.

DETAILED DESCRIPTION:
-Randomized trial with two arms: arm 1: information is delivered by a team (physician and nurse) arm 2: information is delivered by the physician alone

-During the different meetings of the study: at day 1, at day 3, weekly and in case of deterioration of the patient condition.

The other days, family information is delivered as usually in both arms.

ELIGIBILITY:
Inclusion Criteria:

1. patient : adult, 1 relative at minimum, mechanically ventilated at least 48 hours; and
2. family : french-speaking, adult;

Exclusion Criteria:

* Conflict, organ donor, refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Families of patients hospitalized in ICU.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Family satisfaction assessed by qualitative approach | Patient's ICU discharge day (up to 3 months after Day 1)

SECONDARY OUTCOMES:
Healthcaregivers' satifaction assessed by qualitative approach | End of the study (up to 2 years)

OTHER OUTCOMES:
Family PTSD | 3 months after patient's ICU discharge (up to 6 months after Day 1)
Family HADS | 3 months after patient's ICU discharge (up to 6 months after Day 1)
Family peri-traumatic dissociation | Patient's ICU discharge (up to 3 months after Day 1)

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph - Service de Réanimation Polyvalente, Paris, France